CLINICAL TRIAL: NCT00322738
Title: Time to Infection With Malaria Parasites in Adults
Brief Title: Time to Infection With Malaria Parasites
Status: Completed | Type: Observational
Sponsor: National Institute of Allergy and Infectious Diseases (NIAID) (NIH)
Other Study IDs: 05-0067
Record Dates: First submitted 2006-05-04; First posted 2006-05-08 (Estimated); Last update posted 2019-02-01 (Actual); Status verified 2011-11

CONDITIONS: Plasmodium Falciparum Malaria
Keywords: malaria, Plasmodium falciparum, Gambia, larvicides, vector
MeSH Terms: conditions — Malaria, Falciparum; Malaria

STUDY DESIGN:
Time Perspective: Prospective

SUMMARY:
This study will attempt to find out what effect mosquito insecticides have on the transmission of malaria in The Gambia. Eight hundred healthy men and women, aged 18 to 40 years, living in selected villages east of Farafenni town in The Gambia, West Africa will be screened for parasites. About 552 of these people are expected to be free of malaria and will form the study group. These people will participate in the study for 7 months and will be checked for the malaria-causing parasite every two weeks by finger prick blood sample.

DETAILED DESCRIPTION:
Malaria remains one of the world's greatest childhood killers and is a substantial obstacle to social and economic development in the tropics. The overwhelming bulk of the world's malaria burden rests upon the population of sub-Saharan Africa because of the unique coincidence of expanding human populations, weak health systems, the world's most effective vector mosquito species and environmental conditions ideal for transmission. At the start of the new millennium malaria is still deeply entrenched in Africa and effective malaria control is under threat from the inexorable spread of parasite strains resistant to antimalarial drugs and the emergence of mosquitoes resistant to the pyrethroid insecticides used to impregnate bednets. Larval control may offer a new alternative for effective control. Mosquito larval control strategies (environmental management and larviciding) have historically been shown to be successful in reducing the abundance of mosquitoes. This study plans to apply a larvicide in an effort to control malaria and reduce the burden of malaria. While it is abundantly clear that this product will kill mosquito larvae in the laboratory and in the field, it is not certain that doing so will reduce the burden of malaria for the human population. Briefly, the steps involved include survival and development of immature mosquito stages, emergence of adult mosquitoes, blood feeding by those mosquitoes, acquisition and development of malaria parasites by adult mosquitoes and transmission of parasites to susceptible humans. The objective of this pilot study is to evaluate the use of the time-to-infection end point as a measure of malaria transmission in The Gambia, while mosquito larvicides are used to control malaria vectors. The main outcomes of this study are (1) the proportion of adults with detectable parasitemia (Plasmodium falciparum) that is a binary variable and (2) time-to-infection with malaria parasites that will be treated as a continuous variable. This experimental design takes place over 7 months. The target sample size is 800 adults (aged 18-40 years, approximately half will be women and half men) living in 50 villages east of Farafenni town in The Gambia, West Africa. It is estimated that 552 of the adults will have no detectable parasites in their blood at the beginning of the transmission season (June). These parasite negative individuals will be followed either for the duration of the transmission season (June through November) or until they become positive for parasites.

ELIGIBILITY:
Inclusion Criteria:

1. Healthy adults living in the selected villages who consent to join the study,
2. between the ages of 18 to 40 years old, and
3. free of clinical signs or symptoms of illness at recruitment.

Exclusion Criteria:

1. Adults who do not consent to join the study,
2. sick men and women (i.e., have clinical signs or symptoms of illness),
3. men and women 41 years or older, or
4. children.

Ages: 18 Years to 40 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 2558
Dates: Start 2006-06-07; Primary Completion 2008-03-31 (Actual); Study Completion 2009-03-31 (Actual)

CONTACTS AND LOCATIONS:
Locations (1):
- Medical Research Council's Laboratories, Fajara, The Gambia